CLINICAL TRIAL: NCT01704170
Title: A Feasibility Study: An Evaluation of Renal Denervation Using Externally Focused Therapeutic Ultrasound on Patients With Refractory Hypertension
Brief Title: Feasibility Study to Evaluate Renal Denervation Using Focused Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kona Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM12-001
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Denervation Using Externally Focused Ultrasound Therapy (Experimental)
  Interventions: Device: Kona Externally Focused Ultrasound Therapy

INTERVENTIONS:
Device: Kona Externally Focused Ultrasound Therapy

SUMMARY:
This study is a prospective, multi-center trial wherein each included subject will receive the experimental externally focused ultrasound renal denervation therapy. It will be conducted on a maximum of fifty patients who meet the inclusion and exclusion criteria and have signed the informed consent form. Safety is the primary endpoint of this study and will be assessed by incidence and evaluation of any serious adverse effects associated with the investigational procedure through the 52-week evaluation. Clinical utility is the secondary endpoint of this study and will be evaluated by assessing pre and post therapy systolic and diastolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject has systolic blood pressure of 160 mmHg in average or greater.
* Subject has refractory, stable hypertension despite being treated with at least three hypertensive drugs.
* Subject has two functioning kidneys, defined as eGFR ≥ 45 ml/min.
* Subject has at least one renal artery on each side which is greater than 4mm.

Exclusion Criteria:

* Subject has hydronephrosis as seen on MRA or ultrasound.
* Subject has renal stenosis greater than 50% based on baseline MRA.
* Subject has a renal stent or other implant in the region.
* Subject has kidney stones which are symptomatic and/or greater than 1cm or in the discretion of the investigator may interfere with treatment.
* Subject has a history of abdominal surgery within the past six months.
* Subject has heterogeneities in the kidney such as large cysts or tumors which in the discretion of the investigator may interfere with treatment.
* Subject has active pyelonephritis or a history of pyelonephritis which in the discretion of the investigator may interfere with treatment.
* Subject has a history of myocardial infarction, unstable angina pectoris, or cerebrovascular accident within the last six months.
* Subject has hemodynamically significant valvular heart disease.
* Subject has an implantable cardioverter defibrillator, pacemaker, neurostimulator or other device incompatible with MRI.
* Subject has a body weight > 150 kilograms.
* Subject has a target treatment depth > 14 cm.
* Subject is pregnant, nursing or intends to become pregnant during the trial period.
* Subject is currently enrolled in other potentially confounding research.
* Subject has any condition that, at the discretion of the investigator, would preclude participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of Adverse Events through 52 week follow-up | One Year
  Safety will be assessed by incidence and evaluation of any serious adverse effects associated with the investigational procedure through the 52-week evaluation of bilateral treatment. Included in this assessment will be the proportion of subjects with any of the following outcomes: (1) death, or (2) medical morbidity, including but not limited to renal artery aneurysm, stenosis, significant deterioration of renal function, fistulae or ureteral stenosis.

SECONDARY OUTCOMES:
Decrease in Blood Pressure | 12 and 24 weeks post therapy
  Clinical utility will be evaluated by assessing pre and post therapy systolic and diastolic blood pressure.

CONTACTS AND LOCATIONS:
Locations (4):
- Monash Medical Center, Melbourne, Australia
- St. Paul's Hospital, Vancouver, British Columbia, Canada
- Czechia (2):
  - St. Anne's University Hospital, Brno
  - Nemocnice Na Homolee Hospital, Prague